CLINICAL TRIAL: NCT02902549
Title: Real-time Quantitative Optical Perfusion Imaging in Surgery: a Prospective, Observational, In-vivo, Human, Single-center Study
Brief Title: Real-time Quantitative Optical Perfusion Imaging in Surgery
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Quest Medical Imaging (Industry)
Responsible Party: Principal Investigator, S.S. Gisbertz, dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL52377.018.15
Record Dates: First submitted 2016-01-24; First posted 2016-09-16 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Complications of Perfusion
Keywords: Optical Coherence Tomography; Fluorescence Imaging; Sidestream Darkfield Microscopy; Laser Speckle Contrast Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Surgeons are nowadays unable to visualize and quantitatively evaluate microvascularisation in real-time during surgery. Complications due to vascular compromise are a major problem, especially in reconstructive surgery. Poor blood perfusion leads to ischemia and even tissue necrosis. If, however, perfusion and ischemia could be monitored during surgery, then surgeons could change their reconstructive design and the anaesthesiologists could improve perfusion with fluids, inotropes or vasopressors, if necessary. Surgeons therefore need a tool that is able to image in high resolution (microvascularisation), direct, intra-operative, in 3D (to image thrombosis, luminal narrowing or distinct overlaying vessels) and that produces quantitative data to objectify image interpretation.

Optical techniques, based on the interaction of light with tissue, are able to image tissue at high resolution and in real-time. These techniques are FDA-approved and have emerged as powerful diagnostic tools in different departments of medicine, such as ophthalmology for visualizing retina vascularisation and dermatology for skin diagnostics.

In this study, investigators hypothesize that four novel optical technologies: Fluorescence Imaging, Laser Speckle Contrast Imaging, Optical Coherence Tomography and Sidestream Darkfield Microscopy are able to quantitatively image perfusion in real-time during surgery.

DETAILED DESCRIPTION:
Primary objective - Perfusion will be measured with all the techniques focussed on 4 areas; from 'good' to 'decreased' perfusion (biologically)

Fluorescence Imaging (FI): Time to intensity measurements at four sides Laser Speckle Contrast Imaging (LSCI): Perfusion Units Optical Coherence Tomography (OCT): Vessel density & decorrelation time Sidestream Darkfield Microscopy (SDF): Total vessel density, proportion of perfused vessels, perfused vessel density, max flow index, De Backer score, perfusion in mm/sec.

Differences in parameters between the four sites will be statistically be compared.

Secondary objectives

- Relation of parameters to patient outcome in terms of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years - Scheduled for reconstructive surgery with free flap reconstruction or laparoscopic transhiatal and 3-stage transthoracic gastric tube surgery.

Exclusion Criteria:

* Allergic to iodide (indocyanine green)
* Hyper-thyroidism
* Breastfeeding
* No informed consent
* Allergic to ephedrine
* Ischaemic heart disease
* Thyrotoxicosis
* Autonomic thyroid adenomas
* Intraoperative hypertension or tachycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving reconstructive surgical treatment in the Academic Medical Center: 20 patients receiving free flap reconstructive surgery, and 20 patients receiving thoracolaparoscopic esophagectomy with gastric tube reconstruction. Patients will be selected irrespective of medical history, ethnic background or gender, stated that a physician of the department of Biomedical Engineering and Physics is available at time of surgery.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with OCT. | 1 year
  - Perfusion will be imaged with OCT and measured in total vessel density.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in microvascular flow index.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with LSCI. | 1 year
  flux in perfusion units (LSCI)
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with FI. | 1 year
  intensity/time (FI)

SECONDARY OUTCOMES:
Distance of watershed to fundus (GT) or artery to tip (flap) | 1 year
  In the FI images the distance between the end of the right gastroepiploic artery and the fundus, and the distance between the artery entry and tip of the flap can be calculated.
Measurement-time during surgery | 30 minutes
  time in minutes will be calculated during measurements
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with OCT. | 1 year
  - Perfusion will be imaged with OCT and measured in decorrelation time.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in total vessel density.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in perfused vessel density.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in proportion of perfused vessels.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in De Backer Score.
Difference in perfusion between the antrum and fundus (GT) or the artery origin and tip (free flap) measured with SDF. | 1 year
  Perfusion will be imaged with SDF and measured in velocity in mm/sec.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Jansen SM, de Bruin DM, van Berge Henegouwen MI, Strackee SD, Veelo DP, van Leeuwen TG, Gisbertz SS. Can we predict necrosis intra-operatively? Real-time optical quantitative perfusion imaging in surgery: study protocol for a prospective, observational, in vivo pilot study. Pilot Feasibility Stud. 2017 Nov 25;3:65. doi: 10.1186/s40814-017-0204-1. eCollection 2017. PMID 29209513